CLINICAL TRIAL: NCT06066918
Title: The Effect of Preventional Drug Therapy on Pain Regulation Mechanisms Among Spinal Cord Injury Patients Who Have Yet to Develop Central Pain
Brief Title: Prophylactic Pregabalin Treatment Following Spinal Cord Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Loewenstein Hospital (Other)
Responsible Party: Principal Investigator, amiram-catz, Principal Investigator, Loewenstein Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0012-19-LOE
Record Dates: First submitted 2023-09-28; First posted 2023-10-04 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Spinal Cord Injuries; Spinal Cord Diseases
MeSH Terms: conditions — Spinal Cord Injuries; Spinal Cord Diseases | interventions — Pregabalin

STUDY DESIGN:
Intervention Model Description: allocation will be sequential. 2 patients will be in the study group, followed by one patient at the control group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pregabalin (Experimental): Pregabalin 75 mg X2
  Interventions: Drug: Pregabalin 75mg
- No treatment (No Intervention): no treatment

INTERVENTIONS:
Drug: Pregabalin 75mg — Pregabalin 75 mg twice a day
  Other Names: Lyrica
  Arms: Pregabalin

SUMMARY:
Patients arriving to rehabilitation up to 3 months following SCI will be given (study group) or not (control group) Lyrica (75X2). They will be followed for central pain development.

DETAILED DESCRIPTION:
Patients arriving to rehabilitation up to 3 months following SCI will be recruited, if they have not yet developed central pain. Two thirds (the study group) will be treated with Lyrica (Pregabalin75X2) for 3 months. One third (the control group) will not receive preventative treatment. Participants will be followed for central pain development.

ELIGIBILITY:
Inclusion Criteria:

* Up to 3 months following traumatic or non-traumatic SCL
* Ability to give informed consent and cooperate

Exclusion Criteria:

* Pregnancy
* Neurological or other medical conditions that may interfere with sensation
* Neuropathic-like pain before recruitment (described as painful sensation of electric current, burning, numbness, tingling, pricking, or squeezing)
* Being treated with Pregabalin
* Blood creatinine levels >1.2 or creatinine clearance <60
* Sensitivity to lactose

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-07-13 (Actual); Primary Completion 2026-02-05 (Estimated); Study Completion 2026-02-05 (Estimated)

PRIMARY OUTCOMES:
Central pain | 1 year
  development of central pain by interview (yes /no )
McGill Pain Questionnaire | 3 months
  Range 0 -78. higher scores mean worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Amiram Catz, Catz, Principal Investigator — Loewenstein Rehabilitation Hospital
Locations (1):
- Loewenstein Rehabilitation Hospital, Raanana, Israel

DOCUMENTS (1):
  • Study Protocol (2023-02-01): https://cdn.clinicaltrials.gov/large-docs/18/NCT06066918/Prot_000.pdf